CLINICAL TRIAL: NCT00817596
Title: Prometra's Utilization in Mitigating Pain (PUMP)
Acronym: PUMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Flowonix Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G060192
Record Dates: First submitted 2009-01-05; First posted 2009-01-06 (Estimated); Results first posted 2012-07-31 (Estimated); Last update posted 2012-08-17 (Estimated); Status verified 2012-08

CONDITIONS: Intractable Pain
MeSH Terms: conditions — Pain, Intractable | interventions — Infusion Pumps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Infusion Pump (Prometra) — Implantation of pump/catheter for infusion of morphine into the intrathecal space
  Other Names: Prometra

SUMMARY:
Clinical evaluation of the safety and efficacy of the Prometra Programmable Infusion Pump to accurately supply drug to the intrathecal space for the treatment of chronic pain.

DETAILED DESCRIPTION:
Chronic conditions of pain and spasticity are and have been major challenges to traditional medical treatment. Chronic pain and spasticity seriously reduce the quality of life and restrict normal daily activities for many people. The first line of defense is normally oral medications. However, a significant number of these patients require additional or alternative therapy due to the side effects of the oral medications or the intractable nature of the condition.

In 1979, Wand et. al. found that small amounts of morphine, when injected into the sub-arachnoid space, had significant affect in reducing pain. Since that time a number of drug products and infusion pumps have been developed to address this condition. The primary drug used for this purpose in preservative-free morphine sulfate solution which is delivered via an implanted intrathecal catheter. The Prometra Intrathecal Pump System is only the second programmable pump to be used in the treatment of chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* suffering from chronic pain
* 18 years of age or older
* life expectancy >6 months
* failure to respond to less invasive methods
* patient undergone successful morphine trial
* patient agrees with Protocol requirements
* patient considered good subject per clinician

Exclusion Criteria:

* Existing spinal problems that prevent treatment
* systemic infection
* patient is pregnant or breast feeding
* known allergy or sensitivity to materials
* coexisting medical condition that precludes pump usage
* subject requires MRI post procedure
* subject unwilling/unable to comply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2007-01; Primary Completion 2008-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Pain Control Network, Louisville, Kentucky
  - Center for Pain Management, St Louis, Missouri
  - Forsyth Medical Center, Winston-Salem, North Carolina

RESULTS

PARTICIPANT FLOW:
Groups:
- Prometra Intrathecal Pump System: This group was treated with an intrathecal pump implant. Pumps were filled with morphine sulfate. Dosage, concentration, and other programmable parameters were prescribed at the discretion of the physician.
Period: Overall Study
Arm/Group | Prometra Intrathecal Pump System
Started | 110
Completed | 62
Not Completed | 48

BASELINE CHARACTERISTICS:
Arm/Group | Prometra Intrathecal Pump System
Number analyzed (Participants) | 110
Age Continuous [Mean (Standard Deviation); unit: years] | 56 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 59

OUTCOME MEASURES:

1. Primary Outcome: Demonstrate That Prometra Programmable Pump System Accurately and Safely Delivers Medication in the Intrathecal Space, as Programmed.
Description: Accuracy was determined by calculation of the delivered to programmed drug volume (DP) ratio. The DP ratio was calculated as the ratio of delivered drug volume (the volumetrically determined delivered drug volume) to the programmed drug volume (the volume of drug that was programmed to be delivered) summed cumulatively for all fill/refills, including any unscheduled visits per patient.
  The delivered drug volume over all (scheduled and unscheduled) valid fill/refill sessions was summed together per patient as the numerator and the programmed drug volume over all valid fill/refill sessions was summed together per patient as the denominator to provide a per-patient DP ratio.
Time Frame: 6 months - acute study
Population: Sample size was based on previous testing and data from similar devices. With a population of 60 subjects the 90% CI would be 95 ± 7, or 0.88 to 1.02. Therefore, approximately 60 patients with 6-months of data will provide adequate data to demonstrate accuracy, although up to 110 patients may be implanted to account for patient drop-outs.
Measure: Mean (90% Confidence Interval); unit: % of programmed vol. actually delivered
Groups:
- Group 1: Prometra Intrathecal Pump System
Arm/Group | Group 1
Number analyzed (Participants) | 110
% of programmed vol. actually delivered | 97.8 [97.4 to 98.3]

ADVERSE EVENTS:
Time Frame: Up to 3 years and 7 months.
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 11/110
Other Adverse Events (participants affected / at risk) | 110/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=110)
Implant Site Infection (Infections and infestations) | 3 (3)
Diplegia (temporary) (Nervous system disorders) | 1 (1)
Drug Withdrawal Syndrome (General disorders) | 1 (1)
Extradural abscess (Infections and infestations) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Implant Site Cellulitis (Infections and infestations) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Post Lumbar Puncture Syndrome (Injury, poisoning and procedural complications) | 1 (1)
Procedural Pain (Injury, poisoning and procedural complications) | 1 (1)
Surgery to replace pump (Surgical and medical procedures) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=110)
Nausea (Gastrointestinal disorders) | 15 (18)
Vomiting (Gastrointestinal disorders) | 8 (9)
Implant Site Pain (General disorders) | 24 (27)
Implant Site Edema (General disorders) | 11 (15)
Implant Site Erythema (General disorders) | 11 (11)
Pain (General disorders) | 7 (9)
Incision Site Infection (Infections and infestations) | 6 (7)
Procedural Pain (Injury, poisoning and procedural complications) | 37 (39)
Wound secretion (Injury, poisoning and procedural complications) | 9 (13)
Post Lumbar Puncture Syndrome (Injury, poisoning and procedural complications) | 8 (10)
Seroma (Injury, poisoning and procedural complications) | 6 (7)
Headache (Nervous system disorders) | 9 (9)
Surgery (device-related) (Surgical and medical procedures) | 13 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days